CLINICAL TRIAL: NCT05084053
Title: A Phase 3 Study to Evaluate the Efficacy, Safety and Tolerability of TAK-771 for the Treatment of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal Motor Neuropathy (MMN) in Japanese Subjects
Brief Title: A Study of TAK-771 in Japanese Participants With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal Motor Neuropathy (MMN)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-771-3002; jRCT2051210110 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-10-10; First posted 2021-10-19 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP); Multifocal Motor Neuropathy (MMN)
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: TAK-771 for CIDP Participants (Experimental): TAK-771 includes Immune Globulin Infusion (IGI) 10% and Recombinant Human Hyaluronidase (rHuPH20). Participants will receive subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 2, 3, or 4 weeks.
  Interventions: Drug: TAK-771
- Cohort 2: TAK-771 for MMN Participants (Experimental): TAK-771 includes IGI 10% and rHuPH20. Participants will receive subcutaneous infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 2, 3, or 4 weeks.
  Interventions: Drug: TAK-771

INTERVENTIONS:
Drug: TAK-771 — Intervention description; Immune Globulin Infusion (IGI) 10% and Recombinant Human Hyaluronidase (rHuPH20)
  Other Names: Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase

SUMMARY:
The main aim of the study is to check for side effects from TAK-771, and to check how well TAK-771 controls symptoms in Japanese participants with chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) and multifocal motor neuropathy (MMN)

The participants will be treated with TAK-771 for 45 months as a maximum.

There will be many clinic visits. The number of visits will depend on the infusion cycles of study drug (every 2, 3, or 4 weeks).

ELIGIBILITY:
Inclusion criteria

1. Be a Japanese person.
2. The participant is male or female >=18 years old at the time of screening.
3. Participant has a documented diagnosis of definite or probable CIDP (focal atypical CIDP and pure sensory atypical CIDP will be excluded) or definite or probable MMN, as confirmed by a neurologist specializing/experienced in neuromuscular diseases to be consistent with the European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) 2010 criteria.
4. Participant has responded to IgG treatment in the past (partial or complete resolution of neurological symptoms and deficits), and must currently be on stable doses of IVIG treatment within the dose range equivalent to a cumulative monthly dose of 0.4 to 2.4 g/kg BW (inclusive) administered intravenously for at least 12 weeks prior to screening. The dosing interval of intravenous immunoglobulin (IVIG) treatment must be between 2 and 6 weeks (inclusive). Variations in the dosing interval of up to ±7 days or monthly dose amount of up to +or-20% between participant's pre-study IgG infusions are within acceptable limits.
5. CIDP participants only - INCAT disability score between 0 and 7 (inclusive). Participants with INCAT scores of 0, 1 (whether from upper or lower extremities), or 2 (if at least 1 point is from an upper extremity) at screening and/or baseline will be required to have a history of significant disability as defined by an INCAT disability score of 2 (must be exclusively from the lower extremities) or greater documented in the medical record. Participants will be eligible if one of the below eligibility criteria are met:

   1. Screening and Baseline INCAT disability score between 3 and 7 inclusive.
   2. Screening and/or Baseline INCAT disability score of 2 (both points are from lower extremities)
   3. Screening and/or Baseline INCAT disability score of 2 (both points are not from lower extremities) AND has at least a score of 2 or greater documented in the medical record prior to screening. If a score was greater than 2 documented in the medical record prior to screening at least 2 points must be from lower extremities.
   4. Screening and/or Baseline INCAT disability score of 0 or 1 AND has at least a score of 2 or greater (both from lower extremities) documented in the medical record prior to screening, at least 2 points must be from lower extremities.
6. If female of childbearing potential, the participant must have a negative pregnancy test at screening and agree to employ a highly effective contraceptive measure throughout the course of the study and for at least 30 days after the last administration of IP.
7. The participant is willing and able to sign an Informed Consent Form (ICF).
8. The participant is willing and able to comply with the requirements of the protocol.

Exclusion Criteria CIDP patients

1. Participants with focal atypical CIDP or pure sensory atypical CIDP or multifocal acquired demyelinating sensory and motor neuropathy (MADASAM).
2. Participants with any neuropathy of other causes, including:

   1. Hereditary demyelinating neuropathies, such as hereditary sensory and motor neuropathy (HSMN) (Charcot-Marie-Tooth [CMT] disease), and hereditary sensory and autonomic neuropathies (HSANs).
   2. Neuropathies secondary to infections, disorders, or systemic diseases such as Borrelia burgdorferi infection (Lyme disease), diphtheria, systemic lupus erythematosus, POEMS (polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes) syndrome, osteosclerotic myeloma, diabetic and non-diabetic lumbosacral radiculoplexus neuropathy, lymphoma, and amyloidosis.
   3. Multifocal motor neuropathy (MMN).
   4. Drug-, biologic-, chemotherapy-, or toxin-induced peripheral neuropathy. MMN patients
3. Participant with other neuropathies (eg, diabetic, lead, porphyric or vasculitic neuropathy, chronic inflammatory demyelinating polyradiculoneuropathy, Lyme neuroborreliosis, post radiation neuropathy, hereditary neuropathy with liability to pressure palsies, CMT neuropathies, meningeal carcinomatosis).

   CIDP/MMN Patients
4. Participant with immunoglobulin M (IgM) paraproteinemia, including IgM monoclonal gammopathy with high titer antibodies to myelin-associated glycoprotein.
5. Participant with presence of prominent sphincter disturbance.
6. Participant with any central demyelinating disorders such as multiple sclerosis.
7. Participant with any chronic or debilitating disease, or central nervous disorder that causes neurological symptoms or may interfere with assessment of endpoint measures, including (but not limited to) arthritis, stroke, Parkinson's disease, and diabetic peripheral neuropathy.

   (Participants with clinically diagnosed diabetes mellitus who do not have diabetic peripheral neuropathy and who have adequate glycemic control with hemoglobin A1c [HbA1c] level of <7.5% at screening will be eligible for the study, provided the electrodiagnostic criteria are consistent with the diagnosis of a definite or probable CIDP consistent with the EFNS/PNS 2010 criteria and the participant agrees to maintain adequate glycemic control.)
8. Participant with congestive heart failure (New York Heart Association [NYHA] class III/IV), unstable angina, unstable cardiac arrhythmias, or uncontrolled hypertension (defined as diastolic blood pressure >100 mmHg and/or systolic blood pressure >160 mmHg).
9. Participant with a history of deep vein thrombosis or thromboembolic events (eg, cerebrovascular accident, pulmonary embolism) within 12 months prior to screening.
10. Participant with condition(s) which could alter protein catabolism and/or IgG utilization (eg, protein-losing enteropathies, nephrotic syndrome).
11. Participant with a known history of chronic kidney disease, or glomerular filtration rate of <60 mL/min/1.73m^2 estimated based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation at the time of screening.
12. Participant with active malignancy requiring chemotherapy and/or radiotherapy, or history of malignancy with less than 2 years of complete remission prior to screening. Exceptions to this exclusion are: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and stable prostate cancer not requiring treatment.
13. Participant with clinically significant anemia that precludes repeated blood sampling during the study, or hemoglobin (Hgb) level of <10.0 g/dL at the time of screening.
14. Participant with a known history of hypersensitivity or ARs such as urticaria, breathing difficulty, severe hypotension, or anaphylaxis following administration of human blood products such as human IgG, albumin, or other blood components.

    (Clinically non-significant skin reactions, as per the investigator's and the sponsor medical monitor's discretion, do not meet this exclusion criterion. Clinically non-significant skin reactions may include local reactions to injection such as injection site's itching, redness, erythema, or swelling.)
15. Participant has a known allergy to hyaluronidase of human (including recombinant human hyaluronidase) or animal origin such as bee or wasp venom.
16. Participant with immunoglobulin A (IgA) deficiency and antibodies against IgA and a history of hypersensitivity.
17. Participant with an abnormal laboratory values at screening meeting any one of the following criteria:

    1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN).
    2. Platelet count <100,000 cells/microL.
    3. Absolute neutrophil count (ANC) <1000 cells/microL.
18. Participant has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAG), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2.
19. Participant has received or is currently receiving treatment with immunomodulatory/immunosuppressive agents within 6 months prior to screening.
20. Participant has received or is currently receiving treatment with any corticosteroids dose within 8 weeks prior to screening, regardless of indication.
21. Participant has undergone PE within 3 months prior to screening.
22. Participant has any disorder or condition that in the investigator's judgment may impede the participant's participation in the study, pose increased risk to the participant, or confound the results of the study.
23. Participant is nursing or intends to begin nursing during the course of the study.
24. Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment, or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
25. Participant is a family member or employee of the investigator.
26. Participants with known acquired or inherited thrombophilic disorders. These will include the specific types of acquired or inherited thrombophilic disorders that could put participants at risk of developing thrombotic events. Examples include a. Hereditary thrombophilia: i. Factor V Leiden mutation. ii. Prothrombin 20210A mutation. iii. Protein C deficiency. iv. Protein S deficiency. v. Anti-thrombin deficiency. b. Acquired thrombophilia: i. Anti-phospholipid antibody syndrome. ii. Activated protein C Resistance acquired. iii. Homocystinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2026-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (23):
- Japan (23):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa Medical Center, Asahikawa, Hokkaido
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - St.Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Higashimatsuyama Municipal Hospital, Higashi-Matsuyama, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokushima University Hospital, Tokushima, Tokushima
  - Tokushima National Hospital, Yoshinogawa, Tokushima
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Toyama University Hospital, Toyama, Toyama
  - Yamaguchi University Hospital, Ube, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/616f8da3eb0e19002afd68f8

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in Japan. A total of 26 participants were enrolled and treated in this study, which consisted of two treatment epochs (Epoch 1 and Epoch 2) with two cohorts: chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) in Cohort 1 and multifocal motor neuropathy (MMN) in Cohort 2.
Pre-assignment Details: The results are presented up to Epoch 2 (6 months), based on the second interim analysis cutoff date (August 20, 2024). The study is ongoing, and participants who have tolerated the treatment well and voluntarily wish to continue TAK-771 administration may remain in Epoch 2 (continued) until the commercial availability of TAK-771. Additional results will be provided upon study completion date.
Groups:
- Epoch 1, Cohort 1 (CIDP): TAK-771: TAK-771 included Immune Globulin Infusion (IGI) 10 percent (%) and Recombinant Human Hyaluronidase (rHuPH20). Participants with CIDP received subcutaneous (SC) infusion of rHuPH20 solution at a dose of 80 units per gram (U/g) immunoglobulin G (IgG) first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3 or 4 weeks for up to 6 months in Epoch 1 or until relapse.
- Epoch 1, Cohort 2 (MMN): TAK-771: TAK-771 included IGI 10% and rHuPH20. Participants with MMN received SC infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3 or 4 weeks for up to 6 months in Epoch 1.
- Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771: TAK-771 included IGI 10% and rHuPH20. Participants with CIDP received SC infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3 or 4 weeks for 6 months in Epoch 2 (6 months). The dose and dosing interval of TAK-771 in the first 6 months of Epoch 2 were fixed as same as those in Epoch 1. At the end of the first 6 months of Epoch 2, the dosing interval of TAK-771 could be adjusted at the discretion of investigator as medically necessary.
- Epoch 2 (6 months), Cohort 2 (MMN): TAK-771: TAK-771 included IGI 10% and rHuPH20. Participants with MMN received SC infusion of rHuPH20 solution at a dose of 80 U/g IgG first, followed by SC infusion of 10% IGI within 10 minutes of completion of the infusion of rHuPH20 solution, every 3 or 4 weeks for 6 months in Epoch 2 (6 months). The dose and dosing interval of TAK-771 in the first 6 months of Epoch 2 were fixed as same as those in Epoch 1. At the end of the first 6 months of Epoch 2, the dosing interval of TAK-771 could be adjusted at the discretion of investigator as medically necessary.
Period: Epoch 1: Up to 6 months
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Started | 19 | 7 | 0 | 0
Treated | 19 | 7 | 0 | 0
Completed | 17 | 7 | 0 | 0
Not Completed | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: Epoch 2: Up to 6 months
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Started | 0 | 0 | 16 (CIDP participants who completed the 6 months of Epoch 1 entered in the Cohort 1 of Epoch 2 (6 months). One participant of Cohort 1 (CIDP) completed Epoch 1 but not entered Epoch 2 (6 months) due to Lack of Efficacy reason.) | 7 (MMN participants who completed the 6 months of Epoch 1 entered in the Cohort 2 of Epoch 2 (6 months).)
Treated | 0 | 0 | 16 | 7
Completed | 0 | 0 | 15 | 7
Not Completed | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all enrolled participants who received TAK-771 at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Total
Number analyzed (Participants) | 19 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (17.27) | 57.4 (15.71) | 55.6 (16.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 11 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 7 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 7 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Epoch 1: Percentage of Participants With CIDP Who Experienced Relapse
Description: Relapse was defined as worsening of functional disability defined as an increase of >=1 point relative to the pre-subcutaneous (pre-SC) treatment baseline score in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability score. The INCAT disability scale was the most widely used assessment tool to measure the functional activity level of participants with CIDP. The INCAT disability scale consisted of upper and lower extremity components, with a maximum of 5 points for the upper extremities (arm disability) and a maximum of 5 points for the lower extremities (leg disability), which were summed for an overall INCAT disability score ranging from 0 to 10 points, where 0 was normal and 10 was severely incapacitated. An adjusted INCAT disability score was the same as the INCAT disability score, with the only exception in the exclusion of changes from 0 (normal) to 1 (minor symptoms) (or vice versa) in upper limb function.
Time Frame: Epoch 1: Baseline up to 6 months
Population: FAS included all enrolled participants who received TAK-771 at least once.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771
Number analyzed (Participants) | 19
percentage of participants | 0 [0.00 to 17.65]

2. Primary Outcome: Epoch 1: Change From Baseline in Maximum Grip Strength in the More Affected Hand in Participants With MMN
Description: The Martin Vigorimeter was used to assess grip strength in both hands. The instrument consisted of a compressible rubber ball that was connected to a manometer. When the rubber ball was squeezed, the force of compression was measured in kilopascal (kPa) ranging from 0 to 160 kPa.
Time Frame: Epoch 1: Baseline up to 6 months
Population: FAS included all enrolled participants who received TAK-771 at least once.
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Epoch 1, Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 7
kPa | -1.1 (12.73)

3. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of investigational product (IP). TEAEs caused in Epoch 1 were defined as AEs that occurred on or after the start of study drug administration, and before the first dose of IP in Epoch 2 (6 months). TEAEs caused in Epoch 2 (6 months) were defined as AEs that began during or after administration of the first dose of IP in Epoch 2 (6 months).
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: Safety analysis set (SAS)included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants | 16 | 7 | 11 | 6

4. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs were defined as any untoward clinical manifestation of signs, symptoms, outcomes (related to IP or not) at any dose: resulted in death, was life-threatening, required inpatient/prolongation of hospitalization, resulted in persistent/significant disability/incapacity, congenital abnormality/birth defect, or any other important medical event.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Related SAEs and TEAEs
Description: Related SAES and TEAEs: that followed a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which possible involvement of the drug cannot be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant medications and concurrent treatments, may also be responsible.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants
  Participants With Related SAEs | 0 | 0 | 0 | 0
  Participants With Related TEAEs | 11 | 5 | 7 | 4

6. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Serious and Non-serious Adverse Reactions (ARs) Plus Suspected ARs
Description: Adverse reactions plus suspected ARs were defined as TEAEs that were considered by the investigator to be related to IP administration, or for which the causality was indeterminate or missing, or that began during infusion of IP or within 72 hours following the end of IP infusion.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants
  Participants with Serious ARs Plus Suspected ARs | 0 | 0 | 0 | 0
  Participants with non-serious ARs Plus Suspected ARs | 12 | 6 | 7 | 4

7. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With SAEs and/or TEAEs Associated With Infusions
Description: Infusion associated SAEs and/or TEAEs were defined as SAEs and/or TEAEs considered to be "infusion-related reactions" by investigators.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants
  Participants with SAEs associated with Infusions | 0 | 0 | 0 | 0
  Participants with TEAEs associated with Infusions | 9 | 5 | 6 | 4

8. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Related SAEs and TEAEs Associated With Infusions
Description: Related SAES and TEAEs: that followed a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which possible involvement of the drug cannot be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant medications and concurrent treatments, may also be responsible. SAEs and TEAEs associated with infusions were the events considered to be "infusion-related reactions" by investigators.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants
  Participants With Related SAEs Associated With Infusions | 0 | 0 | 0 | 0
  Participants With Related TEAEs Associated With Infusions | 9 | 5 | 6 | 4

9. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With TEAEs Temporally Associated With Infusions
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP. TEAEs caused in Epoch 1 were defined as AEs that occurred on or after the start of study drug administration, and before the first dose of IP in Epoch 2 (6 months). TEAEs caused in Epoch 2 (6 months) were defined as AEs that began during or after administration of the first dose of IP in Epoch 2 (6 months). TEAEs temporally associated with infusions defined as AEs occurring during or within 72 hours after completion of an infusion.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants | 12 | 6 | 7 | 4

10. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Serious and Non-serious ARs Plus Suspected ARs Temporally Associated With Infusions
Description: Adverse reactions plus suspected ARs were defined as TEAEs that were considered by the investigator to be related to IP administration, or for which the causality was indeterminate or missing, or that began during infusion of IP or within 72 hours following the end of IP infusion. AEs temporally associated with infusions are defined as AEs occurring during or within 72 hours after completion of an infusion.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants
  Participants with Serious ARs Plus Suspected ARs Temporally Associated with Infusions | 0 | 0 | 0 | 0
  Participants with Non-serious ARs Plus Suspected ARs Temporally Associated with Infusions | 12 | 6 | 7 | 4

11. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Systemic TEAEs Associated With Infusions
Description: Any TEAEs other than local TEAEs were considered a systemic TEAE. Infusion associated TEAEs were defined as TEAE considered to be "infusion-related reactions" by investigators.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants | 3 | 4 | 3 | 2

12. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Treatment-emergent Local Infusion Site Reactions Associated With Infusions
Description: Any reaction with the medical dictionary for regulatory activities (MedDRA) high-level group term (HLGT) of "Administration site reactions" were considered a local infusion site reaction (local TEAE). In addition, any TEAE with Injection Site Reaction Flag = "Yes" was considered a local TEAE. Infusion associated reaction were defined as event considered to be "infusion-related reactions" by investigators.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Participants | 9 | 5 | 5 | 4

13. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped Due to Intolerability and/or AEs
Description: Number of infusions for which the infusion rate was reduced and/or the infusion was interrupted or stopped due to intolerability and/or AEs were reported.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once.
Measure: Number; unit: infusions
Units Other Than Participants: Total Number of Infusions Administered
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 16 | 7
Number analyzed (Total Number of Infusions Administered) | 172 | 65 | 100 | 46
infusions | 2 | 0 | 0 | 1

14. Secondary Outcome: Epoch 1 and 2 (6 Months): Number of Participants With Positive Binding Antibodies, and Positive Neutralizing Antibodies to rHuPH20
Description: Plasma samples for the detection of anti-rHuPH20 binding and neutralizing antibodies were collected. Participants were monitored for the formation of anti-rHuPH20 antibodies using validated anti-rHuPH20 antibody detection assay (also known as the Screening and Confirmatory Binding Assay). Positive antibodies were defined as participants who had anti rHuPH20 antibody titer greater than or equal to (>=) 1:160 at least one time during treatment.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: SAS included all enrolled participants who received TAK-771 administration at least once. Here, "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 19 | 7 | 15 | 7
Participants
  Participants with Positive Antibodies | 2 | 2 | 3 | 2
  Participants with Positive Neutralizing Antibodies: number analyzed (Participants) | 5 | 2 | 6 | 2
  Participants with Positive Neutralizing Antibodies | 0 | 0 | 0 | 0

15. Secondary Outcome: Epoch 1: Percentage of Participants With Clinical Worsening of CIDP
Description: Clinical Worsening of CIDP was defined as a >=8 kPa decrease in hand grip strength in the more affected hand OR >=4 points decrease in Rasch Built Overall Disability Scale (R-ODS) relative to the pre-SC treatment baseline score at 2 consecutive time points. Hand grip strength was measured using the Martin vigorimeter by quantifying air pressure. The R-ODS was a participant self-reported, linearly-weighted overall disability scale that was specifically designed to capture activity and social participation limitations in participants with immune-mediated peripheral neuropathies including CIDP. R-ODS was comprised of 24 items that rate participant's functioning related to a variety of everyday tasks at moment of completion on a scale of 0 to 2 (where 0 indicates it is not possible for the respondent to perform the task and 2 means that task can be performed without difficulty). Total scores range from 0 to 48 and higher scores indicate greater ability to perform daily and social tasks.
Time Frame: Epoch 1: Baseline until end of Epoch 1 or relapse (up to 6 months)
Population: FAS included all enrolled participants who received TAK-771 at least once.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771
Number analyzed (Participants) | 19
percentage of participants | 21.1 [8.51 to 43.33]

16. Secondary Outcome: Epoch 1 and 2 (6 Months): Time to Relapse in Participants With CIDP
Description: Time to relapse was defined as time from the date of the first SC administration of TAK-771 in Epoch 1 or 2 to the date of relapse.
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Population: FAS included all enrolled participants who received TAK-771 at least once.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771
Number analyzed (Participants) | 19 | 16
weeks | NA [NA to NA] — Data for median and 95% confidence interval was not estimable as less than 50% of the participants had event. | NA [NA to NA] — Data for median and 95% confidence interval was not estimable as less than 50% of the participants had event.

17. Secondary Outcome: Epoch 1: Change From Pre-subcutaneous Treatment (Baseline) in R-ODS Total Score in Participants With CIDP
Description: The R-ODS was a participant self-reported, linearly-weighted overall disability scale that was specifically designed to capture activity and social participation limitations in participants with immune-mediated peripheral neuropathies including CIDP. R-ODS was comprised of 24 items that rate participant's functioning related to a variety of everyday tasks at moment of completion on a scale of 0 to 2 (where 0 indicates it is not possible for the respondent to perform the task and 2 means that task can be performed without difficulty). Total scores range from 0 to 48 and higher scores indicate greater ability to perform daily and social tasks.
Time Frame: Epoch 1: Baseline up to 6 months
Population: FAS included all enrolled participants who received TAK-771 at least once. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771
Number analyzed (Participants) | 17
score on scale | 0.1 (3.24)

18. Secondary Outcome: Epoch 1: Change From Pre-subcutaneous Treatment (Baseline) in an Average of Handgrip Strength of Both Hands in Participants With CIDP and MMN
Description: The Martin Vigorimeter was used to assess grip strength in both hands. The instrument consisted of a compressible rubber ball that was connected to a manometer. When the rubber ball was squeezed, the force of compression was measured in kPa ranging from 0 to 160 kPa. Average of grip strength was defined as an average of the two maximum values: maximum of the 3 measurements in the more affected hand and the maximum of the 3 measurements in the less affected hand.
Time Frame: Epoch 1: Baseline up to 6 months
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 17 | 7
kPa | 4.03 (9.749) | -0.36 (10.613)

19. Secondary Outcome: Epoch 1: Change From Pre-subcutaneous Treatment (Baseline) Total Medical Research Council (MRC) Sum Score in Participants With MMN
Description: The MRC sum score served as a measure of muscle strength. The following muscles on each side of the body were examined and the strength of each muscle was rated according to the MRC scale: deltoids, biceps, wrist extensors, iliopsoas, quadriceps, and anterior tibialis. The MRC scale ranged from 0 to 5, where: 0 = no visible contraction; 1 = visible contraction without movement of the limb; 2 = movement of the limb but not against gravity; 3 = movement against gravity over (almost) the full range; 4 = movement against gravity and resistance; and 5 = normal. All scores from both left and right side of the body were summed to obtain the total MRC sum score. The total MRC sum score ranged from 0 (paralysis) to 60 (normal strength) with higher score indication normal strength.
Time Frame: Epoch 1: Baseline up to 6 months
Population: FAS included all enrolled participants who received TAK-771 at least once.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Epoch 1, Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 7
score on scale | -0.3 (3.59)

20. Secondary Outcome: Epoch 1: Number of MMN Participants With Increased Guy's Neurological Disability Scale (GNDS) Score in Upper Limb and Lower Limb Categories
Description: GNDS was a questionnaire which consisted of 12 separate categories (4 to 8 questions per category). The categories included: cognition, mood, vision, speech, swallowing, upper limb function, lower limb function, bladder function, bowel function, sexual function, fatigue, and others. In the current study, only 2 categories; upper limb function and the lower limb function was used for assessment of the disability of participants with MMN. The severity of each subscale (including upper limb and lower limb) was graded from 0 (normal function) to 5 (total loss of function) based according to severity and impact on the individual. The total GNDS score was the sum of the 12 separate scores ranging between 0 and 60 with higher scores indicating loss of function.
Time Frame: Epoch 1: Baseline up to 6 months
Population: FAS included all enrolled participants who received TAK-771 at least once.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1, Cohort 2 (MMN): TAK-771
Number analyzed (Participants) | 7
Participants
  Participants with increased GNDS score in Upper Limb | 1 [lower limit 1.25]
  Participants with Increased GNDS Score in Lower Limb | 0 [lower limit 1.57]

ADVERSE EVENTS:
Time Frame: Epoch 1: Baseline up to 6 months; Epoch 2: Up to 6 months post-Epoch 1
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Epoch 1, Cohort 1 (CIDP): TAK-771 | Epoch 1, Cohort 2 (MMN): TAK-771 | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/7 | 0/16 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/7 | 0/16 | 0/7
Other Adverse Events (participants affected / at risk) | 16/19 | 7/7 | 11/16 | 6/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1, Cohort 1 (CIDP): TAK-771 (N=19) | Epoch 1, Cohort 2 (MMN): TAK-771 (N=7) | Epoch 2 (6 months), Cohort 1 (CIDP): TAK-771 (N=16) | Epoch 2 (6 months), Cohort 2 (MMN): TAK-771 (N=7)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Administration site erythema (General disorders and administration site conditions) | 1 | 1 | 0 | 1
Administration site extravasation (General disorders and administration site conditions) | 2 | 0 | 2 | 0
Administration site haemorrhage (General disorders and administration site conditions) | 0 | 0 | 0 | 1
Administration site pain (General disorders and administration site conditions) | 2 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Feeling hot (General disorders and administration site conditions) | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 1 | 4 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Infusion site discharge (General disorders and administration site conditions) | 1 | 0 | 0 | 0
Infusion site erythema (General disorders and administration site conditions) | 0 | 1 | 0 | 2
Infusion site pain (General disorders and administration site conditions) | 0 | 1 | 0 | 0
Injection site erythema (General disorders and administration site conditions) | 8 | 2 | 4 | 0
Injection site oedema (General disorders and administration site conditions) | 0 | 0 | 1 | 0
Injection site pain (General disorders and administration site conditions) | 0 | 1 | 0 | 0
Injection site pruritus (General disorders and administration site conditions) | 3 | 0 | 1 | 0
Injection site swelling (General disorders and administration site conditions) | 2 | 1 | 1 | 0
Injection site warmth (General disorders and administration site conditions) | 1 | 1 | 0 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Localised oedema (General disorders and administration site conditions) | 1 | 0 | 1 | 0
Malaise (General disorders and administration site conditions) | 1 | 0 | 0 | 0
Multifocal motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders and administration site conditions) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 1
Pyrexia (General disorders and administration site conditions) | 0 | 1 | 2 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT05084053/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05084053/SAP_001.pdf